CLINICAL TRIAL: NCT03324503
Title: A Multicenter, Open-Label Study to Estimate the Effect Sizes of HRCT Endpoints in Response to GLUCOCORTICOID Induction Therapy in Subjects With Pulmonary Sarcoidosis
Brief Title: A Study to Estimate the Effect Sizes of HRCT Endpoints in Response to Glucocorticoid Induction Therapy in Subjects With Pulmonary Sarcoidosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NDS-CP-001; U1111-1201-4544 (Other: WHO); 2017-002001-34 (EudraCT Number)
Record Dates: First submitted 2017-10-12; First posted 2017-10-27 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Sarcoidosis, Pulmonary
Keywords: Pulmonary Sarcoidosis; HRCT; Glucocorticoid; Prednisone; FRI; Prednisolone
MeSH Terms: conditions — Sarcoidosis, Pulmonary | interventions — Glucocorticoids; Prednisone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glucocorticoid ≥ 30 mg/day (Experimental): ≥ 30 mg/day prednisone or prednisolone as per local clinical practice of sarcoidosis initial induction therapy will be taken orally preferably before, during, or immediately after meals or with food or milk, at approximately the same time of day for 8 weeks.
  Interventions: Drug: Glucocorticoid (prednisone or prednisolone)

INTERVENTIONS:
Drug: Glucocorticoid (prednisone or prednisolone) — ≥ 30 mg/day prednisone or prednisolone taken orally as per local clinical practice of sarcoidosis initial induction therapy
  Other Names: prednisone or prednisolone

SUMMARY:
This is a multicenter, single-arm, unblinded/open-label study of the effect size of HRCT endpoints in response to glucocorticoid induction therapy in subjects with a diagnosis of pulmonary sarcoidosis who have not received glucocorticoid as initial sarcoidosis therapy (≥ 20 mg/day prednisone or prednisolone) or other sarcoidosis therapy for at least 3 months prior to enrollment. This study will enroll a total of approximately 24 subjects.

DETAILED DESCRIPTION:
Optimal development of novel treatments for sarcoidosis requires clinical study endpoints that efficiently reflect changes in disease activity over short treatment durations. Such endpoints enable preliminary assessment of candidate drug efficacy in small studies - prior to exposing large cohorts to experimental compounds in pursuit of registrational data.

This study will accordingly investigate the ways that certain HRCT-based functional respiratory imaging (FRI) measures can serve as more quantitative and sensitive endpoints compared to pulmonary function tests to measure drug effect in a short duration small sample size study in patients with pulmonary sarcoidosis. The study is designed to minimize impact on sarcoid care that the patient would have otherwise received. Glucocorticoid (≥ 30 mg/day prednisone or prednisolone) as per local clinical practice of sarcoidosis initial induction therapy will be taken orally in this study. The glucocorticoid dose may be modified depending on ongoing assessment as a part of standard local clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject are male or female ≥ 18 and ≤ 65 years of age, inclusive, at the time of signing the informed consent form (ICF).
2. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
4. Subject has not received glucocorticoid as initial sarcoidosis therapy (≥ 20 mg/day prednisone or prednisolone) or other sarcoidosis therapy for at least 3 months or 5 PK half-lives, whichever is longer, prior to enrollment.
5. Subjects have a diagnosis of pulmonary sarcoidosis:

   1. According to the American Thoracic Society/European Respiratory Society/World Association of Sarcoidosis and other Granulomatous Disorders (ATS/ERS/WASOG) statement, supported by clinical presentation and biopsy-proven noncaseating granulomatous inflammation with no alternative cause of the granulomas;
   2. With radiographic stage II or III disease;
   3. With dyspnea (MRC grade ≥ 1);
   4. With an FVC of ≥ 45% and ≤ 80% of predicted normal value at screening;
   5. With or without concurrent extra-pulmonary sarcoidosis;
   6. Without clinically significant neurosarcoidosis or cardiac sarcoidosis;
   7. Without history of resistance or refractoriness to glucocorticoid induction therapy.
6. Subject is in good health (except for sarcoidosis) as determined by a physical examination at screening.

   a. Stable and mild syndromes associated with normal ageing, that are not expected to affect safe participation or data interpretation are allowed. Examples include, but are not limited to, systemic hypertension, hypothyroidism, prostatic hypertrophy, etc.
7. Contraception Requirements:

   Must comply with the following acceptable forms of contraception. All FCBP1 must use one of the approved contraceptive options as described below while participating in the study and for at least 28 days after the last study visit.

   At the time of study entry, and at any time during the study when a FCBP's contraceptive measures or ability to become pregnant changes, the Investigator will educate the subject regarding contraception options and the correct and consistent use of effective contraceptive methods in order to successfully prevent pregnancy.

   All FCBP must have a negative pregnancy test at screening and on Days 1, 3 and 5. All FCBP subjects who engage in activity in which conception is possible must use one of the approved contraceptive options described below:

   Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy; OR Option 2: Male or female condom (latex condom or non-latex condom NOT made out of natural [animal] membrane [for example, polyurethane]); PLUS one additional barrier(c) contraceptive sponge with spermicide.

   Male subjects (including those who have had a vasectomy) who engage in activity in which conception is possible must use barrier contraception (latex or non-latex condoms NOT made out of natural [animal] membrane [for example, polyurethane]) while on the study and for at least 28 days after the last study visit.
8. Subject has body mass index (BMI) ≥ 17 and ≤ 33 kg/m2 at screening.
9. Subject has clinical laboratory safety test results that are within normal limits or acceptable to the Investigator. Platelet count, absolute neutrophil count, and absolute lymphocyte count must be above the lower limit of normal at screening.
10. Subject is afebrile, with supine systolic blood pressure (BP) ≥ 90 and ≤ 150 mmHg, supine diastolic BP ≥ 50 and ≤ 90 mmHg, and pulse rate ≥ 40 and ≤ 110 bpm at screening.
11. Subject has a normal or clinically acceptable 12-lead ECG at screening.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment. If the result(s) do not satisfy eligibility criteria, subjects will be ineligible to enroll in the study and will be considered a screen failure. Subjects may be re-screened with the approval of the medical monitor:

1. Subject has any significant medical condition, laboratory abnormality, neurological disease or psychiatric illness that would prevent the subject from safely completing the study. Prior evidence of neurological disease must be documented.
2. Subject has any condition that confounds the ability to interpret data from the study.
3. Subject is a pregnant or a nursing female.
4. Subject has received another interventional investigational drug for sarcoidosis within the 3 months prior to screening or 5 PK half-lives, whichever is longer*.
5. Subject has clinically significant lung disease, other than sarcoidosis, such as asthma, chronic obstructive pulmonary disease (COPD), interstitial lung disease (ILD) or lung cancer.

   a. Subject has a history of significant (greater than a wedge) lung resection.
6. Subject is receiving therapy for sarcoidosis associated pulmonary hypertension, or has an indication for such therapy.
7. Subject has uncontrolled diabetes and other contraindications to glucocorticoid therapy.
8. Subject has a history of listeriosis, coccidioidomycosis, histoplasmosis, blastomycosis, treated or untreated tuberculosis or exposure to individuals with tuberculosis.
9. Subject is an active smoker or has > 10 pack-year smoking history. Previous smokers must have discontinued smoking for at least 1 year.
10. Subject is unable to perform any study-related procedure or maneuver.
11. Subject has had any biologic anti-tumor necrosis factor (anti-TNF) therapy within the previous year.
12. Subject has active infection requiring treatment within 30 days prior to screening*.
13. Subject has a positive QuantiFERON-TB Gold tuberculosis test.

    a. In case of an indeterminate result, the test may be repeated once. The repeat result must be negative to permit entry into the study.
14. Subject has active fungal infection (other than candidiasis of the urinary tract*) or active infection with hepatitis B or hepatitis C or a history of either HCV infection or chronic HBV infection.
15. Subject has a history of congenital and/or acquired immunodeficiencies (eg, common variable immunodeficiency, HIV, etc.).
16. Subject has aspartate transaminase (AST), alanine aminotransferase (ALT) or total bilirubin > 2 x the upper limit of normal at screening (unless the increase is considered to be due to sarcoidosis by the Investigator and/or Sponsor's medical monitor).
17. Subject has a serum creatinine level > 1.8 mg/dL (> 159.12 μmol/L)
18. Subject has clinically significant organic heart disease (eg, congestive heart failure), myocardial infarction requiring initiation or change in medical treatment within six months prior to screening.
19. Subject has QTcF of > 450 milliseconds or findings on electrocardiogram (ECG) at screening (eg, an arrhythmia, heart block, etc.) that suggest either significant cardiac sarcoidosis or significant risk of cardiac adverse event over the duration of this study.
20. Subject has a history of malignancy within 5 years (except basal cell carcinoma of the skin that is surgically cured, remote history of cancer now considered cured or positive pap smear with subsequent negative follow-up).
21. Subject is expecting to have elective surgery in the time interval between screening and 10 weeks after the last study visit if the surgery would be expected to confound evaluation of study endpoints or AE assessment.

    * Candidate subjects having these conditions may be re-evaluated upon resolution and entered into the study if all other criteria are met.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in high-resolution computed tomography (HRCT) | Up to approximately 8 weeks
  Is defined as measurements of lobar volumes total lung capacity (TLC) in response to glucocorticoid induction therapy in subjects with pulmonary sarcoidosis.

CONTACTS AND LOCATIONS:
Overall Officials: Gopal Krishna, PhD, Study Director — Celgene
Locations (20):
- United States (10):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins University School of Medicine - Baltimore, Baltimore, Maryland
  - Pulmonary and Critical Care Medicine-Washington University School of Medicine, St Louis, Missouri
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic - Taussig Cancer Institute, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - MultiCare Institute for Research and Innovation, Tacoma, Washington
- Netherlands (3):
  - Catharina Ziekenhuis, Eindhoven
  - Erasmus University Medical Center, Rotterdam
  - Onderzoekscentrum longziekten Zutphen, Zutphen
- United Kingdom (7):
  - University College London Hospitals NHS Foundation Trust - University College Hospital, London
  - Richmond Pharmacology, London
  - Imperial College London - Hammersmith Hospital Campus, London
  - University Hospital of South Manchester NHS Foundation Trust -Wythenshawe Hospital - North West Lung, Manchester
  - Oxford University Hospitals NHS Trust- Churchill Hospital-Oxford Centre for Respiratory Medicine, Oxford
  - Southmead Hospital, Westbury-on-Trym/ Bristol
  - The Royal Wolverhampton Hospitals NHS Trust - Newcross Hospital, Wolverhampton